CLINICAL TRIAL: NCT03830073
Title: Assessment of the Different Etiological and Susceptibility Markers in Patients With Pancreatitis: Investigating IG4, Cytomegalovirus, Coxsackie- Virus, Genetic Polymorphism of Vitamin D Receptor Gene
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham I El-mahdy, Principal Investigator, Assiut University
Other Study IDs: Autoimmune pancreatitis
Record Dates: First submitted 2019-02-02; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Acute Pancreatitis
Keywords: Cytomegalovirus; Coxsackie- virus; Vitamin D receptor gene; IG4; Autoimmune pancreatitis
MeSH Terms: conditions — Pancreatitis; Coxsackievirus Infections; Autoimmune Pancreatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I:: Seventy patients with pancreatitis
  Interventions: Genetic: Measurement of VDR genetic polymorphism
- Group II:: Thirty healthy controls
  Interventions: Genetic: Measurement of VDR genetic polymorphism

INTERVENTIONS:
Genetic: Measurement of VDR genetic polymorphism — VDR genetic polymorphism will be measured by RFLP and correlated with viral, autoimmune markers.

SUMMARY:
Acute pancreatitis (AP) is a multifactorial disease. AP represents a significant number of hospital admissions. Most of the patients are admitted in an acute setting. Early identification of its etiology is an essential step toward the rational approach, both for its implications in the immediate therapy and the prevention of recurrence. Although often obvious, the etiological workup of acute pancreatitis can be challenging.

DETAILED DESCRIPTION:
Acute pancreatitis is the most common pancreatic disorder. Although acute pancreatitis is a benign disease, it often progresses to a serious state, and mortality is still high. Autoimmune pancreatitis (AIP) was first used to describe cases of pancreatitis with narrowing of the pancreatic duct, enlargement of the pancreas, hyper-γ-globulinaemia, and antinuclear antibody (ANA) positivity serologically by indirect immunofluorescence (IIF). The main differential diagnosis is pancreatic cancer, which can be ruled out through radiological, serological, and histological investigations.

Cytomegalovirus (CMV) is a common viral pathogen in humans. It is a lytic virus that causes a cytopathic effect in vitro and in vivo. Seroprevalence for CMV worldwide ranges from 60%-100% but the severity of illness varies. Primary CMV may be asymptomatic or may cause a mild and self-limiting mononucleosis-like syndrome. The self-limiting course of CMV infection typically includes fever, malaise, splenomegaly, mild hepatomegaly, small increases in serum transaminase activity, and variable elevation of serum alkaline phosphatase. CMV infection can cause severe hepatitis, meningitis, encephalitis, myelitis, colitis, pancreatitis and pneumonitis. Coxsackie-B virus can also cause acute pancreatitis.

VDR are also expressed on pancreatic Ɓ cells, and may play an essential role in maintaining normal insulin levels in accordance to glucose concentrations and to maintain glucose tolerance. Because vitamin D acts through VDR, their impairment or reduced functionality, e.g., as a result of polymorphisms occurring in the VDR gene, may have a crucial impact on the balance in the vitamin D concentration in the circulation, and the final metabolite activity throughout the body.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of acute pancreatitis.
* Patients of age 20 years or more who are willing to participate in the study and give their consent for same.

Exclusion Criteria:

* with a history of severe liver disease,
* sepsis
* Chest disease.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Acute pancreatitis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-20 (Estimated)

PRIMARY OUTCOMES:
The mean difference of single nucleotide polymorphism of VDR between pancreatitis patients and healthy controls | Baseline
  Single nucleotide polymorphism of VDR mean difference will be measured by restriction fragment length polymorphism.

REFERENCES:
- [Background] Cieslinska A, Kostyra E, Fiedorowicz E, Snarska J, Kordulewska N, Kiper K, Savelkoul HFJ. Single Nucleotide Polymorphisms in the Vitamin D Receptor Gene (VDR) May Have an Impact on Acute Pancreatitis (AP) Development: A Prospective Study in Populations of AP Patients and Alcohol-Abuse Controls. Int J Mol Sci. 2018 Jun 29;19(7):1919. doi: 10.3390/ijms19071919. PMID 29966312
- [Background] Chan A, Bazerbachi F, Hanson B, Alraies MC, Duran-Nelson A. Cytomegalovirus hepatitis and pancreatitis in the immunocompetent. Ochsner J. 2014 Summer;14(2):295-9. PMID 24940147
- [Background] Shimizu K, Tahara J, Takayama Y, Akao J, Ajihara T, Nagao K, Shiratori K, Tokushige K. Assessment of the Rate of Decrease in Serum IgG4 Level of Autoimmune Pancreatitis Patients in Response to Initial Steroid Therapy as a Predictor of Subsequent Relapse. Pancreas. 2016 Oct;45(9):1341-6. doi: 10.1097/MPA.0000000000000633. PMID 27171510
- [Background] Ozsvar Z, Deak J, Pap A. Possible role of Coxsackie-B virus infection in pancreatitis. Int J Pancreatol. 1992 Apr;11(2):105-8. doi: 10.1007/BF02925981. PMID 1318913